CLINICAL TRIAL: NCT06999005
Title: Minimally Invasive Protocols for the Treatment and Control of Caries Lesions in Children and Adolescents:A Multicenter Longitudinal Interventional Study
Brief Title: Minimally Invasive Protocols for the Treatment and Control of Caries Lesions in Children and Adolescents
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 100YEARMOLAR
Record Dates: First submitted 2025-05-14; First posted 2025-05-31 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Dental Atraumatic Restorative Treatment

STUDY DESIGN:
Intervention Model Description: This multicenter randomized clinical trial uses a parallel assignment model. After an initial screening of 50,000 children aged 6 to 12 years, approximately 2,500 children with active dental caries lesions will be assigned to one of four treatment arms according to lesion severity and subsequently randomized within the appropriate group. Each participant will receive only one of the four interventions and will be followed for 24 months, with evaluations every three months.
Masking Description: This is an open-label study due to the visible and procedural nature of the dental interventions performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Preventive Varnish Application (Protocol 1) (Experimental): Children with no visible carious lesions or early non-cavitated enamel lesions (ICDAS 0 to 2) will receive a single application of Duraphat® fluoride varnish (Colgate®) on first permanent molars and permanent incisors. The varnish will be applied using cotton swabs, following drying of the surfaces. This protocol aims to provide preventive sealing and will be reapplied every three months.
  Interventions: Procedure: Fluoride Varnish Application (Preventive Protocol)
- Active White Spot Lesion Treatment (Protocol 2) (Experimental): Children diagnosed with active enamel caries lesions (ICDAS 1 to 3) will receive Duraphat® fluoride varnish (Colgate®) in four weekly sessions to promote lesion arrest and remineralization. After lesion inactivation, quarterly reapplications will be performed. For first molars and incisors without lesions but still erupting (with gingival operculum), quarterly varnish applications will also be provided.
  Interventions: Procedure: Fluoride Varnish for Active Enamel Lesions
- ART Sealant Application (Protocol 3) (Experimental): Children with occlusal lesions classified as ICDAS 3 or at high risk of caries will receive ART sealants (Atraumatic Restorative Treatment) using high-viscosity glass ionomer cement. The protocol includes professional cleaning, relative isolation, placement of the material, finger pressure sealing, and final fluoride varnish application. Quarterly evaluations and varnish reapplications will be conducted.
  Interventions: Procedure: Atraumatic Restorative Treatment (ART) Sealant
- Atraumatic Restorative Treatment (Protocol 4) (Experimental): Children with dentin-level carious lesions (ICDAS 4 to 6) and pulpal vitality will receive cavity cleaning with cotton pellets and caries removal using manual excavators and PapacarieDUO® gel. The cavity will be restored with high-viscosity glass ionomer cement using finger pressure technique. Fluoride varnish will be applied afterward. Quarterly follow-ups will include clinical evaluation and retreatment if necessary.
  Interventions: Procedure: Atraumatic Restorative Treatment (ART)

INTERVENTIONS:
Procedure: Fluoride Varnish Application (Preventive Protocol) — Single application of Duraphat® fluoride varnish on permanent molars and incisors, repeated every 3 months.
  Arms: Preventive Varnish Application (Protocol 1)
Procedure: Fluoride Varnish for Active Enamel Lesions — Weekly fluoride varnish applications for 4 weeks, followed by quarterly maintenance applications.
  Arms: Active White Spot Lesion Treatment (Protocol 2)
Procedure: Atraumatic Restorative Treatment (ART) Sealant — Sealant placement with high-viscosity glass ionomer using the ART technique, with quarterly fluoride varnish.
  Arms: ART Sealant Application (Protocol 3)
Procedure: Atraumatic Restorative Treatment (ART) — Manual caries removal and cavity restoration with glass ionomer cement, followed by fluoride varnish every 3 months.
  Arms: Atraumatic Restorative Treatment (Protocol 4)

SUMMARY:
This multicenter longitudinal interventional study aims to evaluate the effectiveness of four minimally invasive protocols for the prevention and control of dental caries in children and adolescents. In the first phase, approximately 50,000 children aged 6 to 12 years from five Brazilian cities will undergo dental screening and receive preventive oral health interventions. In the second phase, 2,500 children diagnosed with active caries will be treated with different interventions, depending on lesion severity. All participants will be followed up every three months for 24 months.

DETAILED DESCRIPTION:
This study is a multicenter longitudinal interventional trial coordinated by the Brazilian Society of Pediatric Dentistry (ABOPED) in five Brazilian cities: Santos, Ponta Grossa, Brasília, Fortaleza, and Belém. The aim is to assess the effectiveness of four evidence-based minimally invasive protocols for preventing and managing dental caries in children and adolescents, and to propose a replicable public health model for pediatric oral care.

In the first phase, approximately 50,000 children aged 6-12 years will undergo dental screening using the International Caries Detection and Assessment System (ICDAS). All children will receive health literacy activities, oral hygiene instructions, toothbrushes, fluoride toothpaste (1,100 ppm), and a single application of fluoride varnish (Duraphat®) to permanent molars and incisors.

Children identified with active caries lesions (ICDAS 1-6) will be considered for the second phase. A total of 2,500 participants will be selected and allocated to one of the following four intervention protocols based on clinical diagnosis:

Protocol 1: Single application of fluoride varnish for prevention. Protocol 2: Four weekly applications of fluoride varnish for active white spot lesions, followed by quarterly applications.

Protocol 3: High-viscosity glass ionomer ART sealants (for ICDAS 3), with quarterly fluoride varnish.

Protocol 4: Conventional atraumatic restorative treatment (ART) with glass ionomer (for ICDAS 4-6), plus quarterly fluoride varnish.

Participants will be followed up every three months over a 24-month period.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 6 and 12 years at the time of enrollment
* Presence of at least one erupted permanent first molar
* Diagnosis of active caries lesions classified according to ICDAS (scores 1 to 6)
* Written informed consent signed by a legal guardian and assent signed by the child
* Ability to attend quarterly follow-up visits over a 24-month period

Exclusion Criteria:

* Children requiring endodontic treatment or presenting extensive pulpal involvement
* Presence of systemic diseases or medical conditions that contraindicate dental care
* Known allergy to any material used in the study (fluoride varnish, high-viscosity glass ionomer cement)
* Participation in other clinical dental studies that could interfere with the outcomes

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2500 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Caries Lesion Progression | Baseline, 3, 6, 9, 12, 15, 18, 21, and 24 months
  Evaluation of changes in caries severity using the International Caries Detection and Assessment System (ICDAS) criteria, comparing baseline scores with follow-up assessments. Progression will be considered when there is an increase in the ICDAS score for the same tooth surface, or development of new lesions.

SECONDARY OUTCOMES:
Survival and Integrity of ART Sealants and Restorations | 3, 6, 9, 12, 15, 18, 21, and 24 months
  To evaluate the clinical success and longevity of sealants and restorations placed using the Atraumatic Restorative Treatment (ART) technique, according to the criteria described by Amorim et al. (2014). Each restoration will be scored from 0 (satisfactory) to 9 (not possible to evaluate), with intermediate codes for marginal defects, fractures, or missing restorations.

IPD SHARING:
Plan to Share IPD: No